CLINICAL TRIAL: NCT06040307
Title: Effect of Guiding Sufentanil Administration by Surgical Plethysmographic Index (SPI) Monitoring on Intraoperative Sufentanil Consumption in Patients Having Trauma and Orthopaedic Surgery With a Combination of General and Regional Anesthesia
Brief Title: Guiding Opioid Administration in Patients With Regional Anesthesia
Acronym: GORA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-08
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Nociceptive Pain; Pain, Postoperative; Analgesia; Anesthesia Recovery Period; Opioid Use
Keywords: General Anesthesia; Regional Anesthesia; Analgesia Monitoring
MeSH Terms: conditions — Nociceptive Pain; Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: Participants are assigned to intervention groups by chance
Who Masked: Participant, Outcomes Assessor
Masking Description: Single-blinded to the primary endpoint (intraoperative amount of sufentanil). Participants are not informed about the group assignment (intervention takes place in general anesthesia). The attending anesthesiologists can not be blinded to the group-allocation, because the study involves intervention during the intraoperative treatment. The study is double-blinded regarding the secondary endpoints. Postoperative outcome parameters are assessed by members of the study team. These outcome-assessors are blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPI (Surgical Pleth Index) (Experimental): Opioid administration (sufentanil) guided by by Surgical Pleth Index (SPI) derived from photoplethysmography performed by the device CARESCAPE B650 Patient Monitor from the manufacturer GE (General Electric) Healthcare, Boston, Massachusetts, US. Included in the monitoring system is a software that continuously calculates the SPI from normalized heart rate and pulse wave amplitude derived from finger photoplethysmography. The numerical index ranges between 0 (low sympathetic tone) and 100 (high sympathetic tone). A SPI score between 20 and 50 has been proposed as the target range to guide opioid analgesics. 5 µg Sufentanil will be administered every 5 minutes if SPI score is calculated more than 50.
  Interventions: Procedure: SPI (Surgical Pleth Index)
- Control (No Intervention): Opioid administration (sufentanil) guided according to standard clinical practice of the attending anesthesiologist based upon changes of heart rate, blood pressure, lacrimation, sweating and spontaneous movements of the patient. As an orientation anesthesiologists are advised to administer 5 µg sufentanil if systolic blood pressure is > 140 mmHg or mean blood pressure is > 100 mmHg or heart rate is > 90 /min. If assessed necessary, the anaesthesiologists are allowed to administer higher or lower sufentanil doses up to their discretion.

INTERVENTIONS:
Procedure: SPI (Surgical Pleth Index) — Elective surgery in patients having trauma and orthopedic surgery with a combination of general and regional anesthesia. Opioid titration is guided by SPI during general anesthesia in the experimental arm.
  Arms: SPI (Surgical Pleth Index)

SUMMARY:
General anesthesia is a combination of hypnotic drugs to achieve unconsciousness and opioid analgesics to ensure antinociception. An alternative approach to the intraoperative administration of high potency opioids in order to achieve antinociception during surgery is combining a general anesthesia with a regional anesthesia.

Modern general anesthesia aims to treat nociception induced by surgical stimulation while avoiding an overdose of opioid analgesics and reducing side-effects of opioid administration. Quality and safety of general anesthesia are of major clinical importance and can be improved by adjusting the opioid analgesics to the optimal individual dose needed.

In the current clinical practice, the opioid dosage is usually chosen by clinical judgment. Recently different monitoring devices estimating the effect of nociception during unconsciousness have become commercially available. One of the first commercially available nociception indices was the Surgical Pleth Index (SPI) derived by the CARESCAPE™B650 patient monitor (GE Healthcare).

Until today, it remains unknown whether guiding sufentanil administration by SPI monitoring affects the administered amount of intraoperative and postoperative opioid, immediate postoperative pain in the postanesthesia care unit (PACU) and the quality of postoperative recovery in patients with a combination of general and regional anesthesia. This study aims to investigate whether guiding sufentanil administration by SPI monitoring - compared to routine care - reduces intraoperative sufentanil consumption in patients having trauma and orthopaedic surgery with a combination of general and regional anesthesia.

DETAILED DESCRIPTION:
General anesthesia is a combination of hypnotic drugs and opioid analgesics. Modern general anesthesia aims to treat nociception induced by surgical stimulation while avoiding an overdose of opioid analgesics and reducing side-effects of opioid administration. Underdosing of opioids during surgery can lead to nociception with increased sympathetic tone, elevated levels of stress hormones, unintended patient movement due to nociception as well as increased postoperative pain. On the other hand, overdosing of opioids can lead to negative side effects such as nausea and vomiting, arterial hypotension, immunosuppression, prolonged recovery times, postoperative delirium and an increase in postoperative pain by opioid-induced-hyperalgesia. Anesthesiologists aim for a long-lasting perioperative anesthesia while at the same time trying to reduce the intraoperative and postoperative opioid administration.

An alternative approach to the intraoperative administration of high potency opioids in order to achieve antinociception during surgery is combining a general anesthesia with a regional anesthesia. However, the quality of regional anesthesia cannot be assessed during general anesthesia by the anesthesiologist and patients cannot express pain themselves. Therefore, anesthesiologists tend to administer a certain calculated opioid dose during the operation. If this calculated opioid administration is essential for a sufficient anesthesia or an unnecessary overdose cannot be assessed by the anesthesiologist. Until now there has been no measurement tool that could estimate the effectiveness of regional anesthesia and the absence of nociception during general anesthesia combined with a regional anesthesia.

In recent years, different monitoring devices estimating the effect of nociception during unconsciousness have become commercially available. Such monitoring devices should help physicians to choose the right dose of opioid analgesics during general anesthesia. Among those, the Surgical Pleth Index (SPI) was one of the first commercially available nociception monitoring devices. The SPI is derived by the CARESCAPE™B650 patient monitor (GE Healthcare) and calculates an index value from normalized heart rate and pulse wave amplitude derived by photoplethysmography. The index is presented on a scale from 0 (low sympathetic tone) to 100 (high sympathetic tone). Nevertheless, current literature is inconclusive about the impact of nociception-monitor-guided opioid administration. So far, there is no definitive evidence on anesthesia related outcome parameters like the administered amount of opioid, postoperative short-term recovery, and long-term outcome. Besides, there has been no study evaluating the assessment of the effectiveness of regional anesthesia during general anesthesia by monitoring the intraoperative nociception with the SPI. If the SPI was able to assess nociception, SPI guided opioid administration would prevent unnecessary opioid administration during the operation and reduce the total dose of opioids. Reduction of the intraoperative opioid dose would mean a clinically important benefit for patients against the background of potential risks of opioid administration. Nevertheless, it remains unknown whether guiding sufentanil administration by SPI monitoring effects the administered amount of intraoperative and postoperative opioid, immediate postoperative pain in the postanesthesia care unit (PACU) and the quality of postoperative recovery in patients with a combination of general and regional anesthesia.

This prospective, randomized controlled trial aims to investigate whether guiding sufentanil administration by SPI monitoring - compared to routine care - reduces intraoperative sufentanil consumption in patients having trauma and orthopaedic surgery with a combination of general and regional anesthesia. The hypothesis tested in the present study is that in patients having trauma and orthopaedic surgery with a combination of general and regional anesthesia guiding sufentanil administration of sufentanil guided by SPI monitoring reduces intraoperative sufentanil consumption compared to routine care.

ELIGIBILITY:
Inclusion Criteria:

* Patients having elective trauma or orthopaedic surgery with a combination of general and regional anaesthesia

Exclusion Criteria:

* Preexisting therapy with beta-blockers, cardiac glycosides or pacemakers
* Cardiac arrhythmia (atrial fibrillation, atrioventricular block > I°)
* Intraoperative treatment with ketamine, beta blockers, beta-adrenergic agonists or clonidine
* Serious peripheral or cardiac autonomic neuropathy
* Inability to specify the postoperative pain level
* Postoperative treatment in an Intensive Care Unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Intraoperative Sufentanil Consumption | 1 day
  Compares the amount of intraoperative opioid administration (sufentanil) per minute of general anesthesia and per kg bodyweight between groups.

SECONDARY OUTCOMES:
Highest postoperative pain level at the PACU | 1 day
  Postoperative pain level measured with the highest score in Numeric Rating Scale (NRS) at the postanesthesia care unit (PACU) with a minimum of 0 and a maximum of 10 values. Higher scores mean a worse outcome.
Median postoperative pain level at the PACU | 1 day
  Postoperative pain level measured with the median score in Numeric Rating Scale (NRS) at the postanesthesia care unit (PACU) with a minimum of 0 and a maximum of 10 values. Higher scores mean a worse outcome.
Incidence of moderate to severe postoperative pain | 1 day
  Incidence of moderate to severe postoperative pain (NRS 4-10) at the postanesthesia care unit (PACU)
Postoperative opioids | 1 day
  Postoperative administered amount of opioids in morphine equivalents (mg) at the postanesthesia care unit (PACU)
PONV | 1 day
  Incidence of postoperative nausea and vomiting (PONV) at the postanesthesia care unit (PACU)
PACU stay | 1 day
  Length of stay at the postanesthesia care unit (PACU) (min) until patients reach fit-for-discharge status
Pain after 24 hours | 2 days
  Postoperative pain level at rest measured with the Numeric Rating Scale (NRS) 24 hours after the operation on the ward with a minimum of 0 and a maximum of 10 values. Higher scores mean a worse outcome.
Quality-of-Recovery (QoR-15) | 2 days
  Quality of postoperative recovery measured with the Quality-of-Recovery (QoR-15) Score 24 hours after the operation on the ward with a minimum of 0 and a maximum of 150 values. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Nitzschke, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Department of Anesthesiology; Center of Anesthesiology and Intensive Care Medicine, Hamburg Eppendorf University Medical Center, Hamburg, Germany

REFERENCES:
- [Derived] Koschmieder KC, Pinnschmidt HO, Borst LS, Greiwe G, Kainz E, Fischer M, Nitzschke R. Opioid administration guided by Surgical Pleth Index in patients with a combination of general and regional anaesthesia during trauma and orthopaedic surgery: a double-blind, randomised controlled trial. J Clin Monit Comput. 2025 Oct 3. doi: 10.1007/s10877-025-01363-2. Online ahead of print. PMID 41042488